CLINICAL TRIAL: NCT04035512
Title: The "Expressive Writing" as Psychological Intervention in Bariatric Population. Prospective Longitudinal Multi Centric Study
Brief Title: The Expressive Writing in Bariatric Surgery
Acronym: EWinBSP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Roma La Sapienza (Other)
Collaborators: University College London Hospitals (Other)
Responsible Party: Principal Investigator, Gianfranco Silecchia, Full Professor of Surgery, University of Roma La Sapienza
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 267116L
Record Dates: First submitted 2019-07-17; First posted 2019-07-29 (Actual); Last update posted 2019-07-29 (Actual); Status verified 2019-07

CONDITIONS: Bariatric Surgery Candidate
Keywords: Bariatric surgery; Expressive writing; Obesity; Alexithymia; Adherence
MeSH Terms: conditions — Obesity; Affective Symptoms

STUDY DESIGN:
Intervention Model Description: The sample will be divided into two group, in a randomized way. The expressive writing group that will perform the writing task and the control group that will not perform the writing task. The study includes two measurements, pre-operatively (T0) and 3 months after surgery (T1)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Expressive writing (Experimental): The expressive writing group will perform the writing task, for 3 consecutive days, 20 minutes each day
  Interventions: Other: Expressive writing
- Control group (No Intervention): Any intervention

INTERVENTIONS:
Other: Expressive writing — The procedure for the writing group will be as follow:
  on day 1 the researcher will call the participant at designed time and will provide a brief introduction to the writing task. Participant will be asked to go in a quiet place in their house where they would have no interruptions but can still be close to the phone. Next, participants were given standardized instructions. Then participants will ask to start writing immediately after hanging up the phone and to write for 20 minutes. The researcher will call the participants after 20 minutes. The procedure for the second and third writing days will be identical.
  The above method was previously tested by Zakowski et al., 2004.
  Arms: Expressive writing

SUMMARY:
The aim of the present study is to test the efficacy of a psychological intervention focused on the expressive writing on the weight loss and adherence, 3 months after surgery in obese population undergoing to bariatric surgery. The sample will be divided into two groups: the expressive writing group that will perform the psychological intervention focused on expressive writing, and the control group that will not perform the psychological intervention. The assignment to the two groups will be randomized. The randomization will be carried out leaving each participant free to blindly choose one of the two sealed envelopes containing the writing instruction sheet and an empty sheet, respectively.

All participants will complete psychometric questionnaires 3 days before surgery (T0) and 3 months (T1) after surgery in order to test the predicted variation on the chosen outcome in a very early stage after surgery. In order to assess the adherence level with a non self - report measure, the serum levels of 25(OH)D, B12, sideraemia and iron at T1 will be collected. Moreover, the adherence to follow up visits (surgical, nutritional and psychological) at 1 and 3 months will be assessed.

The main hypothesis is that those patients undergoing expressive writing would have a greater early Excess Weight Loss % (EWL%), lower level of psychological impairment and higher level of adherence to treatment 3 months after surgery, compare to those patients who are not undergoing expressive writing.

DETAILED DESCRIPTION:
Obesity is a multifactorial disease characterized by genetic, social, cultural and psychological factors. Its complex nature requires a multidisciplinary intervention in order to guarantee an optimal outcome. Currently, laparoscopic bariatric surgery represents the gold standard intervention to treat morbid obesity and related comorbidities, as well as to improve quality of life. The expected Excess Weight Loss (%EWL) after the most popular bariatric procedures ranges between 60% and 70%, respectively at 1 and 2 years after surgery. However, literature shows that more than 30% of bariatric patients do not reach the expected weight loss and up to one third regain substantial weight in the long term period. Several studies showed correlation between post-surgery weight loss or %EWL and personality disorders, eating disorders, mood disorders and anxiety disorder. Also childhood traumatic experiences, that could be associated to the development of obesity, had a role in weight loss after surgery and in affecting emotional regulation. Recent studies also showed the role of emotional regulation and in particular as the difficulty in identifying and describing emotions, known as "alexithymia", was associated respectively to lower %Total Weight Loss at 3 and 6 months after gastric bypass and at 12 months after laparoscopic sleeve gastrectomy.

Considering the influence of alexithymia on people living with obesity seeking a weight loss program, it is conceivable that an intervention focused on emotional state could improve outcome after surgery in term of weight loss.

The expressive writing is a form of writing therapy developed primarily by James W. Pennebaker in the late 1980s consisting of writing about stressful and difficult experience for 15-20 min for 3-5 consecutive days, including one's thoughts and feelings. The expressive writing allows people to express and process emotions, feelings, and thoughts related to the life events and consequent changes and this may favor a mental reorganization of the negative events, a greater expression and regulation of the emotions related to them. This intervention could provoke social, emotional, and consequently, psychophysical changes as is showed in patients with chronic diseases and cancer. It is conceivable that the externalization and the processing of the traumatic events linked to the disease, can favor an improvement of the ability of express emotions and the reduction of the negative thoughts associated.

Recruitment: all patients, considered eligible after a multidisciplinary assessment, will be contacted to request participation in the study. Those who accepted the participation, will be randomized in two groups: the expressive writing group that will perform the psychological intervention focused on expressive writing, and the control group that will not perform the psychological intervention. The randomization will be carried out leaving each participant free to blindly choose one of the two sealed envelopes containing the writing instruction sheet and an empty sheet, respectively. Then all the participants of both groups will complete the informed consent and the questionnaires 3 days before surgery (T0).

According to the randomized recruitment all patients of the expressive writing group will be scheduled for 3 consecutive days (20 minutes each day) on which they will complete the writing task. The procedure for the writing group will be as follow:

on day 1 the researcher will call the participant at designed time and will provide a brief introduction to the writing task. Participant will be asked to go a quiet place in their house where they would have no interruptions but can still be close to the phone. Next, participants were given standardized instructions. Then participants will ask to start writing immediately after hanging up the phone and to write for 20 minutes. The researcher will call the participants after 20 minutes. The procedure for the second and third writing days will be identical.

The above method was previously tested by Zakowski et al., 2004. The control group (no expressive writing) will just complete the above mentioned questionnaires.

Both groups will fill the same questionnaires also at 3 months follow up (T1). In order to assess the adherence level with a non self - report measure, the serum levels of 25(OH)D, B12, sideraemia and iron at T1 will be collected according to the blood analysis provided for the hospital protocol of bariatric surgery.

Moreover, the adherence to follow up visits (surgical and nutritional) at 1 and 3 months will be assessed.

The weight measures at T0, and T1 will be collected in order to test the EWL% reached in both groups.

The present study has been approved by the Ethics Committee of the Department of Dynamic and Clinical Psychology "Sapienza" University of Rome on April 3rd, 2019.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria will follow the European Guidelines on Metabolic and Bariatric Surgery (Fried et al., 2014):

  * With BMI ≥ 40 kg/m2, with BMI 35-40 kg/m2 with co-morbidities in which surgically induced weight loss is expected to improve the disorder
  * declared eligible for pre-operative psychological assessment.

Exclusion Criteria:

* presence of a psychiatric disorder or drug/ alcohol abuse
* cognitive impairment
* level of education less than primary school
* revisional surgery.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 136 (Estimated)
Dates: Start 2019-08-01 (Estimated); Primary Completion 2020-08-01 (Estimated); Study Completion 2020-08-01 (Estimated)

PRIMARY OUTCOMES:
Excess Weight Loss (%EWL) | 3 month
  Those patients undergoing expressive writing would have a greater early Excess Weight Loss % (EWL%)
Emotional Regulation (Toronto Alexithymia Scale) | 3 month
  The TAS-20 is a self-administered questionnaire, consisting of 20 items. The scale ranges between 20 to 100 and it allows to identify alexithymic (> 60), not alexithymic (< 51) and probably alexithymic patients (51-60).We expect that those patients undergoing expressive writing would have a lower score (<51) compared to control group patients.
Adherence (Visual Analogue Scale) | 3 month
  The VAS asks individuals to mark a line at the point along a continuum showing how much of each drug they have taken in the past 6 months from 0% to 100% where 0% means you have taken no drug/s in the past 6 months, 50% means you have taken half of your drug/s in the past 6 months and 100% means you have taken all of your drug/s in the past 6 months. After surgery it will be used also to assess the adherence to nutritional supplements provided by the bariatric protocol. We expect that those patients undergoing expressive writing would have a higher level of adherence to treatment on VAS score (>90).

CONTACTS AND LOCATIONS:
Overall Officials: Gianfranco Silecchia, Principal Investigator — University of Roma La Sapienza

IPD SHARING:
Plan to Share IPD: Yes
The personal data will be managed only by the two PhD students involved in this research.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: From the recruitment till 4 years after it ends.
Access Criteria: The data will be managed by the two PhD students involved in the study. All data will be inserted in a an excel database of a University laptop protected from a password. Then, the PhD students will analyze all the data whit an Univariate analysis of variance (ANOVA) on repeated measures in order to test both the difference between the expressive writing group vs control group and the Italian sample vs English sample to verify the hypothesized differences between the groups. Furthermore, correlational models (Pearson r) and predictive models (multivariate regression models) will be performed to verify the associations between the psychological variables, the levels of adherence to treatment and the EWL% reached. To each participant will be assigned a numerical code, in order to guarantee the anonymity.

REFERENCES:
- [Background] Lai C, Aceto P, Petrucci I, Castelnuovo G, Callari C, Giustacchini P, Sollazzi L, Mingrone G, Bellantone R, Raffaelli M. The influence of preoperative psychological factors on weight loss after bariatric surgery: A preliminary report. J Health Psychol. 2019 Mar;24(4):518-525. doi: 10.1177/1359105316677750. Epub 2016 Nov 16. PMID 27852888
- [Background] Paone E, Pierro L, Damico A, Aceto P, Campanile FC, Silecchia G, Lai C. Alexithymia and weight loss in obese patients underwent laparoscopic sleeve gastrectomy. Eat Weight Disord. 2019 Feb;24(1):129-134. doi: 10.1007/s40519-017-0381-1. Epub 2017 Mar 28. PMID 28353096
- [Background] Altamura M, Porcelli P, Fairfield B, Malerba S, Carnevale R, Balzotti A, Rossi G, Vendemiale G, Bellomo A. Alexithymia Predicts Attrition and Outcome in Weight-Loss Obesity Treatment. Front Psychol. 2018 Dec 4;9:2432. doi: 10.3389/fpsyg.2018.02432. eCollection 2018. PMID 30564177
- [Background] Calia R, Lai C, Aceto P, Luciani M, Camardese G, Lai S, Fantozzi C, Pietroni V, Salerno MP, Spagnoletti G, Pedroso JA, Romagnoli J, Citterio F. Emotional self-efficacy and alexithymia may affect compliance, renal function and quality of life in kidney transplant recipients: results from a preliminary cross-sectional study. Physiol Behav. 2015 Apr 1;142:152-4. doi: 10.1016/j.physbeh.2015.02.018. Epub 2015 Feb 11. PMID 25680476
- [Background] Pennebaker JW, Beall SK. Confronting a traumatic event: toward an understanding of inhibition and disease. J Abnorm Psychol. 1986 Aug;95(3):274-81. doi: 10.1037//0021-843x.95.3.274. No abstract available. PMID 3745650
- [Background] Norman SA, Lumley MA, Dooley JA, Diamond MP. For whom does it work? Moderators of the effects of written emotional disclosure in a randomized trial among women with chronic pelvic pain. Psychosom Med. 2004 Mar-Apr;66(2):174-83. doi: 10.1097/01.psy.0000116979.77753.74. PMID 15039501
- [Background] Gallo I, Garrino L, Di Monte V. [The use of expressive writing in the course of care for cancer patients to reduce emotional distress: analysis of the literature]. Prof Inferm. 2015 Jan-Mar;68(1):29-36. doi: 10.7429/pi.2015.681029. Italian. PMID 25837613
- [Background] Fried M, Yumuk V, Oppert JM, Scopinaro N, Torres A, Weiner R, Yashkov Y, Fruhbeck G. [Interdisciplinary European guidelines on metabolic and bariatric surgery]. Rozhl Chir. 2014 Jul;93(7):366-78. Czech. PMID 25263472
- [Background] Figura A, Ahnis A, Stengel A, Hofmann T, Elbelt U, Ordemann J, Rose M. Determinants of Weight Loss following Laparoscopic Sleeve Gastrectomy: The Role of Psychological Burden, Coping Style, and Motivation to Undergo Surgery. J Obes. 2015;2015:626010. doi: 10.1155/2015/626010. Epub 2015 Nov 15. PMID 26649192
- [Background] Taylor GJ. Alexithymia: concept, measurement, and implications for treatment. Am J Psychiatry. 1984 Jun;141(6):725-32. doi: 10.1176/ajp.141.6.725. PMID 6375397
- [Background] Lodhia NA, Rosas US, Moore M, Glaseroff A, Azagury D, Rivas H, Morton JM. Do adverse childhood experiences affect surgical weight loss outcomes? J Gastrointest Surg. 2015 Jun;19(6):993-8. doi: 10.1007/s11605-015-2810-7. Epub 2015 Apr 2. PMID 25832488
- [Background] Palmisano GL, Innamorati M, Vanderlinden J. Life adverse experiences in relation with obesity and binge eating disorder: A systematic review. J Behav Addict. 2016 Mar;5(1):11-31. doi: 10.1556/2006.5.2016.018. PMID 28092189
- [Background] Semanscin-Doerr DA, Windover A, Ashton K, Heinberg LJ. Mood disorders in laparoscopic sleeve gastrectomy patients: does it affect early weight loss? Surg Obes Relat Dis. 2010 Mar 4;6(2):191-6. doi: 10.1016/j.soard.2009.11.017. Epub 2010 Jan 1. PMID 20189470
- [Background] Livhits M, Mercado C, Yermilov I, Parikh JA, Dutson E, Mehran A, Ko CY, Gibbons MM. Preoperative predictors of weight loss following bariatric surgery: systematic review. Obes Surg. 2012 Jan;22(1):70-89. doi: 10.1007/s11695-011-0472-4. PMID 21833817
- [Background] Karlsson J, Taft C, Ryden A, Sjostrom L, Sullivan M. Ten-year trends in health-related quality of life after surgical and conventional treatment for severe obesity: the SOS intervention study. Int J Obes (Lond). 2007 Aug;31(8):1248-61. doi: 10.1038/sj.ijo.0803573. Epub 2007 Mar 13. PMID 17356530
- [Background] Capoccia D, Coccia F, Guarisco G, Testa M, Rendina R, Abbatini F, Silecchia G, Leonetti F. Long-term Metabolic Effects of Laparoscopic Sleeve Gastrectomy. Obes Surg. 2018 Aug;28(8):2289-2296. doi: 10.1007/s11695-018-3153-8. PMID 29497961
- [Background] Zakowski SG, Ramati A, Morton C, Johnson P, Flanigan R. Written emotional disclosure buffers the effects of social constraints on distress among cancer patients. Health Psychol. 2004 Nov;23(6):555-63. doi: 10.1037/0278-6133.23.6.555. PMID 15546223